CLINICAL TRIAL: NCT00109395
Title: A Randomized Controlled Trial Comparing Lorazepam With Midazolam for Sedation of Mechanically Ventilated Pediatric Patients
Brief Title: Lorazepam Sedation for Critically Ill Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Emmes Company, LLC (Industry)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HHSN275200403367C (contract)
Record Dates: First submitted 2005-04-27; First posted 2005-04-28 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Critical Illness
Keywords: Lorazepam; Midazolam; Best Pharmaceuticals for Children Act; Critically ill; pediatrics; mechanical ventilation; sedation
MeSH Terms: conditions — Critical Illness | interventions — Lorazepam; Midazolam

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lorazepam Intermittent bolus (Active Comparator): lorazepam administered by intermittent bolus
  Interventions: Drug: Lorazepam
- lorazepam continuous infusion (Active Comparator): lorazepam administered by continuous infusion
  Interventions: Drug: Lorazepam CI
- midazolam continous infusion (Active Comparator): midazolam administered by continous infusion
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Lorazepam — Intravenous dosage forms, administered at dose and frequency per protocol in order to achieve adequate sedation as measured by the Comfort score
  Other Names: Ativan
  Arms: Lorazepam Intermittent bolus
Drug: Midazolam — Intravenous dosage forms, administered at dose and frequency per protocol in order to achieve adequate sedation as measured by the Comfort score
  Other Names: Versed
  Arms: midazolam continous infusion
Drug: Lorazepam CI — Intravenous dosage forms, administered at dose and frequency per protocol in order to achieve adequate sedation as measured by the Comfort score
  Other Names: Ativan
  Arms: lorazepam continuous infusion

SUMMARY:
This clinical trial is being performed under the Best Pharmaceuticals for Children Act, signed into law in 2002 in order to improve pediatric labeling for off-patent drugs. The purpose of this study is to make sure that lorazepam, when given to children who are very sick in the Intensive Care Unit and who are on a breathing machine, is safe and works as well as a drug called midazolam. Midazolam is already approved by the FDA for this use, but lorazepam is not, even though both drugs are commonly used for sedation.

DETAILED DESCRIPTION:
Lorazepam is used clinically for sedation of mechanically ventilated children, but has not been approved by the FDA for this indication in children. The purpose of this study, in response to the Written Request by FDA, is to determine the safety, efficacy, and dosage required for lorazepam compared with midazolam, which is approved by FDA for children for this indication.

Study participants must be children who are critically ill and receiving mechanical ventilation who require sedation. Participants will be randomized to lorazepam (intermittent bolus or continuous infusion) or midazolam (continuous infusion). Sedation will be monitored using the COMFORT score. Blood will be drawn to measure lorazepam/midazolam plasma concentrations, and to measure the plasma concentrations of excipients (benzyl alcohol and glycols) in patients receiving lorazepam.

ELIGIBILITY:
Inclusion Criteria:

* Males or females from full term birth (at least 38 weeks post conceptual age) through 18 years
* Patients must be intubated and mechanically ventilated in the PICU less than or equal to 24 hr
* Patients in whom the use of neuromuscular blocking agents would normally NOT be expected to be used.
* Patient's parent or guardian has signed a consent form prior to initiation of study procedures
* Patients with cardiac, renal, or hepatic dysfunction will be actively sought

Exclusion Criteria:

* Life expectancy < 48 hr
* Expected duration of sedation < 48 hr
* Patient with history of hypersensitivity to any component of lorazepam, midazolam, fentanyl, thiopental
* Females pregnant or breast feeding
* Patient requires sedatives or analgesics other than study drug

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 179 (Actual)
Dates: Start 2004-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Rate of Severe Adverse Events | Minimum 8 hours
  Duration of study participation
Number of bolus doses required to achieve a comfort score of 17 ≤ 26 | minimum of 8 hours
  A measurement of drug efficacy
Drug dose required to maintain a target comfort score of 17 ≤ 26 | Minimum of 8 hours
  Measurement of efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Blumer, MD, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States